CLINICAL TRIAL: NCT05386030
Title: A Randomized, Subject- and Evaluator-blinded, Controlled, Non-inferiority Multicenter, Parallel Group Comparison Study to Evaluate Effectiveness and Safety of Saypha® VOLUME Lidocaine for Midface Augmentation to Correct Volume Deficit
Brief Title: Saypha® VOLUME Lidocaine for Midface Augmentation
Acronym: VOLIDO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-301-201417
Record Dates: First submitted 2021-05-11; First posted 2022-05-23 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-08

CONDITIONS: Moderate to Severe Midface Volume Deficit

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- saypha® VOLUME Lidocaine (Experimental): For injection, either a needle (27G ½'') or cannula (25G 1½") may be used. Randomization will be stratified by injection equipment in a 1:1 ratio.
  The volume administered is at the discretion of the treating investigator and depends on the severity of the midface volume deficit to be corrected. However, the maximum volume (left and right side of the midface together) must not exceed 10 mL in total per treatment (initial and repeat-treatment) or 20 mL per 60 kg (130 lbs) body mass per year.
  Interventions: Combination Product: saypha® VOLUME Lidocaine
- Juvéderm® Voluma™ XC (Active Comparator): For injection, either a needle (27G ½'') or cannula (25G 1½") may be used. Randomization will be stratified by injection equipment in a 1:1 ratio.
  The volume administered is at the discretion of the treating investigator and depends on the severity of the midface volume deficit to be corrected. However, the maximum volume (left and right side of the midface together) must not exceed 10 mL in total per treatment (initial and repeat-treatment) or 20 mL per 60 kg (130 lbs) body mass per year.
  Interventions: Combination Product: Juvéderm® Voluma™ XC

INTERVENTIONS:
Combination Product: saypha® VOLUME Lidocaine — Crosslinked hyaluronic acid (HA) 23 mg/mL + 0.3% lidocaine hydrochloride.
  Arms: saypha® VOLUME Lidocaine
Combination Product: Juvéderm® Voluma™ XC — Crosslinked HA 20 mg/mL + 0.3% lidocaine hydrochloride
  Arms: Juvéderm® Voluma™ XC

SUMMARY:
The clinical investigation is a randomized, subject- and evaluator-blinded, active treatment controlled, multicenter, clinical investigation, to demonstrate the non inferiority of saypha® VOLUME Lidocaine to one of the devices approved for the same indication (Juvéderm® Voluma™ XC).

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, comparator-controlled study. The study took place in the US at 16 sites.

The purpose of the current clinical investigation is to evaluate the effectiveness, safety and long-term safety of saypha® VOLUME Lidocaine for the correction of age-related moderate to severe volume deficit in the midface (augmentation of midface volume deficit), and to demonstrate its non-inferiority to one of the devices approved for the same indication (Juvéderm® Voluma™ XC). In addition, the duration of the aesthetic effect after implantation will be studied.

Approximately 486 subjects in total will be randomized and treated resulting in 437 evaluable subjects for the primary endpoint. Randomization will be in a 2:1 ratio (test device: 324, comparator device: 162).

Each subject will take part in the investigation for up to 92 weeks. The total anticipated duration of the investigation, from the first-subject-first visit to the last-subject-last-visit, is around 114 weeks, based on expected recruitment period of about 22 weeks.

ELIGIBILITY:
Inclusion Criteria: (baseline treatment)

1. Male or female subjects aged 22 - 75 years (inclusive) of age at Screening.
2. Subjects with bilateral, approximately symmetric moderate to severe midface volume deficit (severity scores of 2 or 3 on the 5-point Midface Volume Deficit Severity Scale), as assessed by the blinded investigator at the site.
3. Females of childbearing potential must have a negative urine pregnancy test and must agree to use an effective method of birth control throughout the entire study. Male subjects with female partners of child-bearing potential must agree to use contraception throughout the entire study (surgical sterilization or a physical barrier such as a condom).
4. Healthy skin in the midface area and free of diseases that could interfere in cutaneous aging evaluation.
5. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of entire investigation, including botulinum toxin injection (except glabella or forehead botulinum toxin treatment).
6. Subjects who understand the purpose and conduct of the study and having given written informed consent and are willing and able to attend the study visits as judged by the investigator.

Exclusion Criteria: (baseline treatment)

1. Females, who are pregnant and/or, lactating or planning to become pregnant during the clinical investigation
2. History of severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies
3. History of hypersensitivity to hyaluronic acid preparations, lidocaine or any amide-based anesthetic
4. Tendency to keloid formation and/or hypertrophic scars and/ or have pigment disorders
5. Known human immune deficiency virus-positive individuals
6. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the treatment area
7. Re-current (three times a year over the last year) herpes simplex in the treatment area
8. History or presence of any autoimmune or connective tissue disease, or current treatment with immuno-modulating therapy
9. Uncontrolled (or unstable) Diabetes mellitus or systemic diseases as per investigator discretion
10. Previous facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) and semi-permanent / long-lasting fillers (e.g., poly-L-lactic acid (PLLA), Polymethylmethacrylate (PMMA) filler) in the area of device application and during the entire investigation
11. Implantation of dermal fillers in the treatment area within the preceding 24 months prior to Visit 1 (Screening) and during the entire investigation
12. Subject has received any of the following aesthetic treatments in the midface area: e.g., laser therapy, absorbable and non-absorbable sutures (threads), dermabrasion, mesotherapy, micro-needling and/or botulinum toxin (including treatment of crow´s feet in the outer eye region) within the last 12 months prior to Visit 1, chemical peeling within the last three months prior to Visit 1 or is planning to undergo such procedures during entire investigation.
13. Facial lipolysis, including submental fat treatments, within the previous 12 months prior to Visit 1 (Screening) and during the entire investigation
14. Bariatric surgery within 12 months prior to Visit 1 (Screening) and during the entire investigation
15. History of bleeding disorder and/or use of anticoagulant, antiplatelet, thrombolytic medication, or anti-inflammatory drugs (oral/injectable corticosteroids or non steroidal anti-inflammatory drugs, e.g., Motrin® or Advil®) or other substances known to increase coagulation time (vitamins or herbal supplements, e.g., St. John's Wort, high doses of vitamin E supplements) from ten days pre- to seven days post injection (baseline treatment and touch-up treatment)
16. Planned dental/oral surgery or modification (bridge-work, implants) within four weeks prior to each injection and to a minimum of four weeks post injection baseline treatment and touch-up treatment
17. Beard longer than three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the investigator
18. Subjects who have one of the following assessments during the visual examinations at Visit 2 (Baseline): Snellen visual acuity test worse than 20/40 (with corrective eyewear, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test.
19. Subjects with active COVID-19 infection and subjects with symptoms consistent with COVID-19 infection including any other respiratory symptoms/illnesses within the past 14 days unless tested negative prior to Visit 1 (Screening)
20. Any medical condition prohibiting the inclusion in the study according to the judgment of the treating investigator
21. Previous enrollment in this clinical investigation
22. Current participation in another clinical trial, or treatment with any investigational drug/medical device within 30 days prior to Visit 1 (Screening) or within five half-lives of an investigational drug, whichever is longer and during the entire investigation
23. Midface volume deficit due to a congenital defect, trauma, or abnormalities in facial adipose tissue distribution such as those associated with HIV related lipodystrophy
24. Subjects who experienced weight change for a minimum of 10% over the last 12 months (e.g., post bariatric patients), or subjects who have the intention to change eating habits that result in a weight gain or loss >10% during the entire investigation
25. Any individual whose willingness to volunteer in this clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants).
26. Close affiliation with the investigator (e.g., a close relative, financially dependent on the study site) or subject who is an employee of the sponsor's company or group companies of the sponsor.

Inclusion criteria: (touch-up treatment)

1. Females of childbearing potential must have a negative urine pregnancy test

Exclusion criteria: (touch-up treatment)

1. Occurrence of a related Serious Adverse Event or Adverse Event of Special Interest (i.e., embolic events, with possible, probable, or causal relationship to an intravascular injection of the device, as changes in vision [loss of vision, blurriness, double vision, pain in or around the eye, blindness, blind spots, problems moving the eyes], skin changing color around the eyelids or around the site of injection, other embolic phenomenon, e.g., stroke, skin necrosis, or impending necrosis) during or after the previous injections
2. Subjects who experienced visual changes considered abnormal clinically significant or other serious medical conditions during or after the previous injections
3. Subjects who have one of the following assessments during the visual examinations: Snellen acuity test worse than 20/40 (with corrective eyewear, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test.

Inclusion criteria: (repeat-treatment)

1. Subjects with bilateral, approximately symmetric moderate to severe midface volume deficit (severity scores of 2 or 3 on the 5-point MVDSS), as assessed by the blinded evaluator at the site. The subject does not have to return to his baseline severity to be permitted to receive a repeat-treatment.
2. Subject has completed initial treatment phase up to Visit 9 (SV1) and is willing to attend the study visits of the screening phase for repeat-treatment and repeat-treatment phase
3. Females of childbearing potential must have a negative urine pregnancy test
4. Healthy skin in the midface area and free of diseases that could interfere in cutaneous aging evaluation

Exclusion criteria: (repeat-treatment)

1. Occurrence of a related Serious Adverse Event or Adverse Event of Special Interest (i.e., embolic events with possible, probable, or causal relationship to an intravascular injection of the device, as changes in vision [loss of vision, blurriness, double vision, pain in or around the eye, blindness, blind spots, problems moving the eyes], skin changing color around the eyelids or around the site of injection, other embolic phenomenon, e.g., stroke, skin necrosis, or impending necrosis) during or after the baseline injection and/or touch-up injections
2. Occurrence of a related Adverse Event that occurred during the initial treatment phase, and is ongoing at the time of the repeat treatment (i.e., relationship is classified as "possible", "probable" or "causal relationship"; outcome is "not recovered / resolved", "recovering / resolving", "recovered / resolved with sequelae" or "unknown")
3. Subjects who experienced visual changes considered abnormal clinically significant or other serious medical conditions during or after the baseline or touch-up injections, respectively
4. Subjects who have one of the following assessments during the visual examinations: Snellen acuity test worse than 20/40 (with corrective eyewear, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test
5. Subjects who became pregnant since start of the study or planning to become pregnant during the clinical investigation
6. Known human immune deficiency virus-positive individuals
7. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the treatment area
8. Development of re-current (three times a year over the last year) herpes simplex in the treatment area since study start
9. Development of any autoimmune or connective tissue disease since study start, or current treatment with immuno-modulating therapy
10. Development of uncontrolled (or unstable) diabetes mellitus or systemic diseases since study start as per investigator discretion
11. Facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) and semi-permanent fillers (e.g., poly-L-lactic acid) in the area of device application and during the initial treatment phase of the investigation
12. Implantation of dermal fillers (other than the test and comparator device used in the investigation) in the treatment area during the initial treatment phase of the investigation
13. Subject has received any of the following aesthetic treatments in the midface area: e.g., laser therapy, absorbable and non-absorbable sutures (threads), dermabrasion, mesotherapy, micro-needling and/or botulinum toxin (including treatment of crow´s feet in the outer eye region), or chemical peeling during the initial treatment phase of the investigation or is planning to undergo such procedures during the repeat-treatment phase of the investigation
14. Facial lipolysis, including submental fat treatments during the initial treatment phase of the investigation
15. Bariatric surgery during the initial treatment phase of the investigation
16. Development of bleeding disorder and/or use of anticoagulant, antiplatelet, thrombolytic medication, or anti-inflammatory drugs (oral/injectable corticosteroids or non steroidal anti-inflammatory drugs, e.g., Motrin® or Advil®) or other substances known to increase coagulation time (vitamins or herbal supplements, e.g., St. John's Wort, high doses of vitamin E supplements) from ten days pre- to seven days post injection (repeat-treatment and touch-up treatment)
17. Planned dental/oral surgery or modification (bridge work, implants) within four weeks prior to the injection and to a minimum of four weeks post injection
18. Any medical condition prohibiting the inclusion for repeat-treatment according to the judgement of the treating investigator
19. Beard longer than three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the investigator
20. Previous enrollment in initial treatment phase of this clinical investigation and early termination, or significant incompliance with the protocol requirements
21. Current or previous treatment with another investigational drug and/or medical device or participation in another clinical study
22. Midface volume deficit due to a trauma, or abnormalities in facial adipose tissue distribution such as those associated with HIV related lipodystrophy
23. Subjects who experienced weight change for a minimum of 10% since study start or subjects who have the intention to change eating habits that result in a weight gain or loss >10% during the entire investigation
24. Subjects with active COVID-19 infection and subjects with symptoms consistent with COVID-19 infection including any other respiratory symptoms/illnesses within the past 14 days unless tested negative prior to Visit RT1

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse S Rafal, MD, Principal Investigator — DermResearchCenter of New York
Locations (16):
- United States (16):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Clinical Testing of Beverly Hills, Encino, California
  - Center for Dermatology Cosmetic & Laser Surgery, Fremont, California
  - Cosmetic Laser Dermatology, San Diego, California
  - About Skin, Greenwood Village, Colorado
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Skin Associates of South Florida, Coral Gables, Florida
  - Meridian Clinical Research, Georgia Plastic Surgery, Savannah, Georgia
  - Chicago Cosmetic, Chicago, Illinois
  - Skin Specialists, Omaha, Nebraska
  - Imagedermatology PC, Montclair, New Jersey
  - Luxurgery, New York, New York
  - DermResearchCenter of NY, Stony Brook, New York
  - Aesthetic Solutions, Chapel Hill, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch Inc. Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 562 enrolled participants, 486 met inclusion criteria and were randomized to treatment.
Groups:
- Saypha® VOLUME Lidocaine: For injection, either a needle (27G ½'') or cannula (25G 1½") may be used. Randomization will be stratified by injection equipment in a 1:1 ratio.
  The volume administered is at the discretion of the treating investigator and depends on the severity of the midface volume deficit to be corrected. However, the maximum volume (left and right side of the midface together) must not exceed 10 mL in total per treatment (initial and repeat-treatment) or 20 mL per 60 kg (130 lbs) body mass per year.
  saypha® VOLUME Lidocaine: Crosslinked hyaluronic acid (HA) 23 mg/mL + 0.3% lidocaine hydrochloride.
- Juvéderm® Voluma™ XC: For injection, either a needle (27G ½'') or cannula (25G 1½") may be used. Randomization will be stratified by injection equipment in a 1:1 ratio.
  The volume administered is at the discretion of the treating investigator and depends on the severity of the midface volume deficit to be corrected. However, the maximum volume (left and right side of the midface together) must not exceed 10 mL in total per treatment (initial and repeat-treatment) or 20 mL per 60 kg (130 lbs) body mass per year.
  Juvéderm® Voluma™ XC: Crosslinked HA 20 mg/mL + 0.3% lidocaine hydrochloride
Period: Overall Study
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Started | 324 | 162
Received Treatment | 322 | 161
Completed | 280 | 143
Not Completed | 44 | 19
Not completed — Death | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 19 | 7
Not completed — Withdrawal by Subject | 20 | 10
Not completed — Eligibility criteria violation | 1 | 1
Not completed — Personal Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population used consists of all randomized subjects who received at least one injection with study medication. Participants were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC | Total
Number analyzed (Participants) | 322 | 161 | 483
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 263 | 132 | 395
  >=65 years | 59 | 29 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.7) | 56.0 (9.5) | 55.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 154 | 457
  Male | 19 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 28 | 96
  Not Hispanic or Latino | 254 | 133 | 387
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 7 | 16
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 20 | 7 | 27
  White | 283 | 140 | 423
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 322 | 161 | 483
Midface Volume Deficit Severity Scale (MVDSS) by the Blinded Evaluator [Count of Participants; unit: Participants]
  0 (none/minimal) | 0 | 0 | 0
  1 (mild) | 0 | 0 | 0
  2 (moderate) | 189 | 99 | 288
  3 (severe) | 133 | 62 | 195
  4 (very severe) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Responders on the 5-point Mid-Face Volume Deficit Severity Scale (MVDSS) at Week 24 - Per Protocol Dataset
Description: The percentage of responders on the 5-point MVDSS (Mid-Face Volume Deficit Severity Scale where 0 means no deficit and 4 means Extreme Deficit) based on the blinded evaluator´s live assessment at Week 24 after last injection of initial treatment phase compared to the pre-treatment score at Baseline visit. Subjects are defined as responders if they are showing an >=1 point improvement in MVDSS at Week 24 relative to baseline.
Time Frame: Week 24
Population: The population used consists of all randomized subjects, who received at least one administration of the test device or the comparator device and who did not have any major protocol deviation affecting the primary effectiveness endpoint. Subjects with missing baseline Mid-Face Volume Deficit Severity Scale (MVDSS) score and / or missing MVDSS score at Week 24 after last injection of the initial treatment phase were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 275 | 139
Participants | 268 | 124
Statistical Analysis 1: Comparison: Saypha® VOLUME Lidocaine vs Juvéderm® Voluma™ XC; Test type: Non-Inferiority — The hypothesis to be tested was: H0: pA-pB ≤ d0 versus H1: pA-pB> d0 where, pA is the response rate for saypha® VOLUME Lidocaine, pB is the response rate for the Comparator, and d0 is the non-inferiority margin set at -10%. The hypothesis was tested based on Farrington-Manning-statistics with a one-sided type I error rate level of 0.025; p < 0.0001, Farrington-Manning test — Confirmatory testing will be performed in a hierarchical ordering: First analysis will be performed on the per protocol dataset, and if the corresponding p-value is below 0.025, the analysis will be performed on the full analysis dataset

2. Primary Outcome: The Percentage of Responders on the 5-point Mid-Face Volume Deficit Severity Scale (MVDSS) at Week 24 - Full Analysis Dataset
Description: The percentage of responders on the 5-point MVDSS (Mid-Face Volume Deficit Severity Scale where 0 means no deficit and 4 means Extreme Deficit) based on the blinded evaluator´s live assessment at Week 24 after last injection of initial treatment phase compared to the pre-treatment score at Baseline visit. Subjects are defined as responders if they are showing an >=1 point improvement in MVDSS at Week 24 relative to baseline. Subjects with missing baseline MVDSS score and / or missing MVDSS score at Week 24 after last injection of the initial treatment phase were imputed as non-responders.
Time Frame: Week 24
Population: The population used consists of all randomized subjects, who received at least one administration of the test device or the comparator device. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
Participants | 283 | 135
Statistical Analysis 1: Comparison: Saypha® VOLUME Lidocaine vs Juvéderm® Voluma™ XC; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Farrington-Manning test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: The Percentage of Responders on the 5-point Mid-Face Volume Deficit Severity Scale (MVDSS) at Weeks 4, 8, 16, 36, and 48 as Rated by the Blinded Evaluator
Description: The percentage of responders on the 5-point MVDSS (Mid-Face Volume Deficit Severity Scale where 0 means no deficit and 4 means Extreme Deficit), based on the blinded evaluator´s live assessment at Weeks 4, 8, 16, 36, and 48 after last injection of initial treatment compared to the score at Baseline. Subjects are defined as responders if they are showing an >=1 point improvement in MVDSS at the respective visit relative to baseline.
Time Frame: Weeks 4, 8, 16, 36, and 48
Population: The population used consists of all randomized subjects, who received at least one administration of the test device or the comparator device and have data available for the respective visit. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
Participants
  Week 4: number analyzed (Participants) | 299 | 154
  Week 4 | 291 | 149
  Week 8: number analyzed (Participants) | 300 | 152
  Week 8 | 294 | 147
  Week 16: number analyzed (Participants) | 295 | 152
  Week 16 | 286 | 147
  Week 36: number analyzed (Participants) | 282 | 144
  Week 36 | 254 | 115
  Week 48: number analyzed (Participants) | 281 | 143
  Week 48 | 203 | 90

4. Secondary Outcome: The Percentage of Responders on the 5-point Mid-Face Volume Deficit Severity Scale (MVDSS) at Weeks 4, 8, 16, 24, 36, and 48 as Rated by the Independent Blinded Photographic Reviewer
Description: The percentage of responders on the 5-point MVDSS (Mid-Face Volume Deficit Severity Scale where 0 means no deficit and 4 means Extreme Deficit), based on the independent blinded photographic reviewer´s assessment by using photographs at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment compared to the score at Baseline. The median of all assessments for the same photograph were taken into account.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: The population used consists of all randomized subjects, who received at least one administration of the test device or the comparator device and who have data available for the respective visit. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
Participants
  Week 4: number analyzed (Participants) | 294 | 148
  Week 4 | 162 | 78
  Week 8: number analyzed (Participants) | 297 | 150
  Week 8 | 173 | 83
  Week 16: number analyzed (Participants) | 290 | 149
  Week 16 | 170 | 85
  Week 24: number analyzed (Participants) | 285 | 147
  Week 24 | 163 | 77
  Week 36: number analyzed (Participants) | 273 | 138
  Week 36 | 156 | 67
  Week 48: number analyzed (Participants) | 270 | 138
  Week 48 | 147 | 67

5. Secondary Outcome: Mean Change in Midface Volume Deficit
Description: Mean change in midface volume deficit measured on the 5-point MVDSS (Mid-Face Volume Deficit Severity Scale where 0 means no deficit and 4 means Extreme Deficit), and based on the blinded evaluator´s live assessment at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment compared to the score at Baseline.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
score on a scale
  Week 4 - Change from Baseline: number analyzed (Participants) | 299 | 154
  Week 4 - Change from Baseline | -1.8 (0.7) | -1.6 (0.8)
  Week 8 - Change from Baseline: number analyzed (Participants) | 300 | 152
  Week 8 - Change from Baseline | -1.8 (0.7) | -1.6 (0.8)
  Week 16 - Change from Baseline: number analyzed (Participants) | 295 | 152
  Week 16 - Change from Baseline | -1.7 (0.7) | -1.5 (0.7)
  Week 24 - Change from Baseline: number analyzed (Participants) | 292 | 151
  Week 24 - Change from Baseline | -1.6 (0.7) | -1.4 (0.8)
  Week 36 - Change from Baseline: number analyzed (Participants) | 282 | 144
  Week 36 - Change from Baseline | -1.4 (0.8) | -1.2 (0.8)
  Week 48 - Change from Baseline: number analyzed (Participants) | 281 | 143
  Week 48 - Change from Baseline | -1.0 (0.8) | -0.9 (0.8)

6. Secondary Outcome: Mean Change in Midface Volume Deficit as Measured by Volumetric Change Measurement
Description: Mean change in midface volume deficit as measured by volumetric change measurement by using 3D digital photographic images at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment compared to Baseline.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: The population used consists of all randomized subjects, who received at least one administration of the test device or the comparator device and who have data available at the respective visit. Participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
cm^3
  Week 4 - Change from Baseline [cm^3]: number analyzed (Participants) | 297 | 150
  Week 4 - Change from Baseline [cm^3] | 8.538 (4.572) | 6.536 (4.163)
  Week 8 - Change from Baseline [cm^3]: number analyzed (Participants) | 299 | 151
  Week 8 - Change from Baseline [cm^3] | 8.236 (4.561) | 6.711 (4.341)
  Week 16 - Change from Baseline [cm^3]: number analyzed (Participants) | 292 | 151
  Week 16 - Change from Baseline [cm^3] | 7.627 (4.612) | 6.115 (4.900)
  Week 24 - Change from Baseline [cm^3]: number analyzed (Participants) | 290 | 149
  Week 24 - Change from Baseline [cm^3] | 7.315 (4.654) | 5.767 (4.793)
  Week 36 - Change from Baseline [cm^3]: number analyzed (Participants) | 281 | 142
  Week 36 - Change from Baseline [cm^3] | 6.781 (4.575) | 4.739 (5.106)
  Week 48 - Change from Baseline [cm^3]: number analyzed (Participants) | 275 | 142
  Week 48 - Change from Baseline [cm^3] | 6.383 (4.836) | 4.690 (5.426)

7. Secondary Outcome: Change in Nasolabial Folds Measurements
Description: Shift from baseline in nasolabial folds measured by the 5-point validated NLF-SRS (Nasolabial Folds Severity Rating Scale, where 0 means no NLF and 4 means Extreme Nasolabial fold) based on the blinded evaluator´s live assessment at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
units on a scale
  Week 4 - Change from Baseline - Left side of the face: number analyzed (Participants) | 299 | 154
  Week 4 - Change from Baseline - Left side of the face | -0.5 (0.8) | -0.5 (0.7)
  Week 4 - Change from Baseline - Right side of the face: number analyzed (Participants) | 299 | 154
  Week 4 - Change from Baseline - Right side of the face | -0.5 (0.8) | -0.5 (0.7)
  Week 8 - Change from Baseline - Left side of the face: number analyzed (Participants) | 300 | 152
  Week 8 - Change from Baseline - Left side of the face | -0.5 (0.8) | -0.5 (0.7)
  Week 8 - Change from Baseline - Right side of the face: number analyzed (Participants) | 300 | 152
  Week 8 - Change from Baseline - Right side of the face | -0.5 (0.9) | -0.5 (0.7)
  Week 16 - Change from Baseline - Left side of the face: number analyzed (Participants) | 295 | 152
  Week 16 - Change from Baseline - Left side of the face | -0.5 (0.8) | -0.5 (0.8)
  Week 16 - Change from Baseline - Right side of the face: number analyzed (Participants) | 295 | 152
  Week 16 - Change from Baseline - Right side of the face | -0.4 (0.8) | -0.5 (0.8)
  Week 24 - Change from Baseline - Left side of the face: number analyzed (Participants) | 292 | 151
  Week 24 - Change from Baseline - Left side of the face | -0.5 (0.8) | -0.5 (0.8)
  Week 24 - Change from Baseline - Right side of the face: number analyzed (Participants) | 292 | 151
  Week 24 - Change from Baseline - Right side of the face | -0.4 (0.8) | -0.5 (0.8)
  Week 36 - Change from Baseline - Left side of the face: number analyzed (Participants) | 282 | 144
  Week 36 - Change from Baseline - Left side of the face | -0.4 (0.8) | -0.4 (0.8)
  Week 36 - Change from Baseline - Right side of the face: number analyzed (Participants) | 282 | 144
  Week 36 - Change from Baseline - Right side of the face | -0.3 (0.8) | -0.4 (0.8)
  Week 48 - Change from Baseline - Left side of the face: number analyzed (Participants) | 281 | 143
  Week 48 - Change from Baseline - Left side of the face | -0.4 (0.7) | -0.3 (0.8)
  Week 48 - Change from Baseline - Right side of the face: number analyzed (Participants) | 281 | 143
  Week 48 - Change from Baseline - Right side of the face | -0.3 (0.8) | -0.2 (0.8)

8. Secondary Outcome: Proportion of Subjects With Global Aesthetic Improvement Based on Modified Global Aesthetic Improvement Scale (GAIS) as Rated by Blinded Evaluator
Description: The percentage of subjects with a global aesthetic improvement over baseline (subjects who have been rated as "much improved" or "improved"), based on the blinded evaluator's assessment at Weeks 4, 8, 16, 24, 36, and 48, after last injection of initial treatment phase using the 5-point modified Global Aesthetic Improvement Scale (GAIS). The blinded evaluators assess aesthetic improvement via photographs comparing baseline photos against the respective study visit week photo with the following possible 5 outcomes: "Much worse", "Worse", "No change", "Improved", "Much improved".
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: The population used consists of all randomized subjects who received at least one injection with study medication and for whom data are available at the respective timepoint. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
Participants
  Week 4: number analyzed (Participants) | 298 | 154
  Week 4 | 292 | 150
  Week 8: number analyzed (Participants) | 300 | 152
  Week 8 | 298 | 149
  Week 16: number analyzed (Participants) | 294 | 152
  Week 16 | 287 | 149
  Week 24: number analyzed (Participants) | 292 | 151
  Week 24 | 283 | 135
  Week 36: number analyzed (Participants) | 282 | 144
  Week 36 | 261 | 126
  Week 48: number analyzed (Participants) | 280 | 143
  Week 48 | 237 | 105

9. Secondary Outcome: Proportion of Subjects With Global Aesthetic Improvement Based on Modified Global Aesthetic Improvement Scale (GAIS) as Rated by Subject
Description: The percentage of subjects with a global aesthetic improvement over baseline (subjects who have been rated as "much improved" or "improved"), based on the subject's assessment at Weeks 4, 8, 16, 24, 36, and 48, after last injection of initial treatment phase using the 5-point modified Global Aesthetic Improvement Scale (GAIS). The subjects assess aesthetic improvement via photographs comparing baseline photos against the respective study visit week photo with the following possible 5 outcomes: "Much worse", "Worse", "No change", "Improved", "Much improved".
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
Participants
  Week 4: number analyzed (Participants) | 299 | 154
  Week 4 | 283 | 146
  Week 8: number analyzed (Participants) | 302 | 152
  Week 8 | 281 | 142
  Week 16: number analyzed (Participants) | 294 | 152
  Week 16 | 269 | 137
  Week 24: number analyzed (Participants) | 292 | 151
  Week 24 | 255 | 125
  Week 36: number analyzed (Participants) | 282 | 144
  Week 36 | 219 | 120
  Week 48: number analyzed (Participants) | 280 | 143
  Week 48 | 213 | 99

10. Secondary Outcome: Satisfaction With Outcome Based on FACE-Q(TM) Assessed by Subjects
Description: The extent of subject's satisfaction with overall treatment outcome at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment phase as assessed by the subject using the Face-Q(TM) Questionnaire "Satisfaction with Outcome". This validated patient reported outcome is based on subject's answers to pre-specified questions with answers ranging as 1="Definitely disagree", 2="Somewhat disagree", 3="Somewhat agree", 4="Definitely agree". The answers are mathematically transferred to one single numerical result between 100 and 0, where 100 reflects the highest possible satisfaction and 0 means the lowest possible satisfaction.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
score on a scale
  Week 4: number analyzed (Participants) | 299 | 154
  Week 4 | 73.2 (20.6) | 72.6 (21.1)
  Week 8: number analyzed (Participants) | 302 | 152
  Week 8 | 72.1 (23.0) | 70.5 (22.7)
  Week 16: number analyzed (Participants) | 295 | 152
  Week 16 | 68.6 (23.1) | 68.7 (21.6)
  Week 24: number analyzed (Participants) | 292 | 151
  Week 24 | 68.2 (23.4) | 68.4 (22.6)
  Week 36: number analyzed (Participants) | 282 | 144
  Week 36 | 63.7 (24.5) | 64.5 (24.7)
  Week 48: number analyzed (Participants) | 281 | 143
  Week 48 | 63.5 (24.3) | 62.1 (24.6)

11. Secondary Outcome: Appearance Appraisal Based on FACE-Q(TM) Assessed by Subjects
Description: The extent of subject's appearance appraisal at Weeks 4, 8, 16, 24, 36, and 48 after last injection of initial treatment phase as assessed by the FACE-Q(TM) questionnaire "Satisfaction with Cheeks" compared to Baseline visit (i.e., change from baseline). This validated patient reported outcome is based on subject's answers to pre-specified questions with answers ranging as 1="Very Dissatisfied", 2="Somewhat Dissatisfied", 3="Somewhat Satisfied", 4="Very Satisfied". The answers are mathematically transferred to one single numerical result between 100 and 0, where 100 reflects the highest possible satisfaction and 0 means the lowest possible satisfaction.
Time Frame: Weeks 4, 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
score on a scale
  Week 4 - Change from Baseline: number analyzed (Participants) | 298 | 154
  Week 4 - Change from Baseline | 47.7 (29.5) | 44.5 (30.0)
  Week 8 - Change from Baseline: number analyzed (Participants) | 301 | 152
  Week 8 - Change from Baseline | 46.9 (28.3) | 40.4 (31.3)
  Week 16 - Change from Baseline: number analyzed (Participants) | 294 | 152
  Week 16 - Change from Baseline | 42.5 (30.4) | 39.1 (30.1)
  Week 24 - Change from Baseline: number analyzed (Participants) | 291 | 151
  Week 24 - Change from Baseline | 40.2 (30.3) | 36.8 (31.4)
  Week 36 - Change from Baseline: number analyzed (Participants) | 281 | 144
  Week 36 - Change from Baseline | 35.4 (30.1) | 32.8 (30.3)
  Week 48 - Change from Baseline: number analyzed (Participants) | 280 | 143
  Week 48 - Change from Baseline | 34.7 (29.3) | 28.7 (30.2)

12. Secondary Outcome: Pain Assessment by Subjects
Description: Assessment of pain associated with the procedure by subjects immediately after injection and about 15, 30, 45 and 60 minutes thereafter for initial treatment at baseline and for touch-up treatment at week 2 (if applicable). Subjects quantified the pain associated with the procedure using a semi-quantitative 11-point Numeric Pain Rating Scale (NPRS): 0 is no pain and 10 is the worst pain you can imagine. Left and right side of the face was assessed separately.
Time Frame: Baseline - Immediately after end of treatment and 15, 30, 45, 60 minutes after end of treatment; Week 2 - Immediately after end of treatment and 15, 30, 45, 60 minutes after end of treatment
Population: The population used consists of all randomized subjects who received at least one injection with study medication and for whom data are available at the respective timepoint and side of face. Participants were analyzed as randomized. Participants who received Lidocaine before the assessment were excluded from the analysis for the respective visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
score on a scale
  Pain assessment immediately after end of treatment - Baseline - Left: number analyzed (Participants) | 308 | 158
  Pain assessment immediately after end of treatment - Baseline - Left | 2.5 (2.3) | 2.3 (2.2)
  Pain assessment immediately after end of treatment - Baseline - Right: number analyzed (Participants) | 307 | 158
  Pain assessment immediately after end of treatment - Baseline - Right | 2.5 (2.2) | 2.3 (2.3)
  Pain assessment 15 minutes after end of treatment - Baseline - Left: number analyzed (Participants) | 308 | 158
  Pain assessment 15 minutes after end of treatment - Baseline - Left | 0.7 (1.2) | 0.8 (1.3)
  Pain assessment 15 minutes after end of treatment - Baseline - Right: number analyzed (Participants) | 308 | 158
  Pain assessment 15 minutes after end of treatment - Baseline - Right | 0.8 (1.3) | 0.8 (1.4)
  Pain assessment 30 minutes after end of treatment - Baseline - Left: number analyzed (Participants) | 308 | 158
  Pain assessment 30 minutes after end of treatment - Baseline - Left | 0.4 (0.8) | 0.6 (1.0)
  Pain assessment 30 minutes after end of treatment - Baseline - Right: number analyzed (Participants) | 308 | 158
  Pain assessment 30 minutes after end of treatment - Baseline - Right | 0.4 (0.8) | 0.6 (1.0)
  Pain assessment 45 minutes after end of treatment - Baseline - Left: number analyzed (Participants) | 308 | 158
  Pain assessment 45 minutes after end of treatment - Baseline - Left | 0.2 (0.6) | 0.4 (0.9)
  Pain assessment 45 minutes after end of treatment - Baseline - Right: number analyzed (Participants) | 308 | 158
  Pain assessment 45 minutes after end of treatment - Baseline - Right | 0.2 (0.6) | 0.4 (0.9)
  Pain assessment 60 minutes after end of treatment - Baseline - Left: number analyzed (Participants) | 308 | 158
  Pain assessment 60 minutes after end of treatment - Baseline - Left | 0.1 (0.4) | 0.2 (0.6)
  Pain assessment 60 minutes after end of treatment - Baseline - Right: number analyzed (Participants) | 308 | 158
  Pain assessment 60 minutes after end of treatment - Baseline - Right | 0.1 (0.4) | 0.2 (0.5)
  Pain assessment immediately after end of treatment - Week 2 - Left: number analyzed (Participants) | 179 | 95
  Pain assessment immediately after end of treatment - Week 2 - Left | 2.0 (2.5) | 1.8 (2.1)
  Pain assessment immediately after end of treatment - Week 2 - Right: number analyzed (Participants) | 185 | 96
  Pain assessment immediately after end of treatment - Week 2 - Right | 1.9 (2.4) | 1.9 (2.1)
  Pain assessment 15 minutes after end of treatment - Week 2 - Left: number analyzed (Participants) | 179 | 95
  Pain assessment 15 minutes after end of treatment - Week 2 - Left | 0.7 (1.4) | 0.6 (1.2)
  Pain assessment 15 minutes after end of treatment - Week 2 - Right: number analyzed (Participants) | 185 | 96
  Pain assessment 15 minutes after end of treatment - Week 2 - Right | 0.6 (1.4) | 0.7 (1.2)
  Pain assessment 30 minutes after end of treatment - Week 2 - Left: number analyzed (Participants) | 179 | 94
  Pain assessment 30 minutes after end of treatment - Week 2 - Left | 0.4 (1.0) | 0.3 (0.8)
  Pain assessment 30 minutes after end of treatment - Week 2 - Right: number analyzed (Participants) | 185 | 95
  Pain assessment 30 minutes after end of treatment - Week 2 - Right | 0.4 (1.0) | 0.3 (0.8)
  Pain assessment 45 minutes after end of treatment - Week 2 - Left: number analyzed (Participants) | 179 | 93
  Pain assessment 45 minutes after end of treatment - Week 2 - Left | 0.2 (0.8) | 0.2 (0.6)
  Pain assessment 45 minutes after end of treatment - Week 2 - Right: number analyzed (Participants) | 185 | 94
  Pain assessment 45 minutes after end of treatment - Week 2 - Right | 0.2 (0.8) | 0.2 (0.6)
  Pain assessment 60 minutes after end of treatment - Week 2 - Left: number analyzed (Participants) | 179 | 93
  Pain assessment 60 minutes after end of treatment - Week 2 - Left | 0.1 (0.7) | 0.1 (0.5)
  Pain assessment 60 minutes after end of treatment - Week 2 - Right: number analyzed (Participants) | 185 | 94
  Pain assessment 60 minutes after end of treatment - Week 2 - Right | 0.1 (0.7) | 0.1 (0.5)

13. Secondary Outcome: Evaluation of Injection Volume
Description: Injection volume required to achieve optimal aesthetic result at each treatment (baseline and touch-up treatment together) measured in mL.
Time Frame: Baseline and Week 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
Number analyzed (Participants) | 322 | 161
mL | 5.163 (2.306) | 4.975 (2.251)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Saypha® VOLUME Lidocaine | Juvéderm® Voluma™ XC
All-Cause Mortality (participants affected / at risk) | 1/322 | 0/161
Serious Adverse Events (participants affected / at risk) | 4/322 | 2/161
Other Adverse Events (participants affected / at risk) | 84/322 | 41/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saypha® VOLUME Lidocaine (N=322) | Juvéderm® Voluma™ XC (N=161)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saypha® VOLUME Lidocaine (N=322) | Juvéderm® Voluma™ XC (N=161)
Vision blurred (Eye disorders) | 8 (8) | 1 (1)
Injection site bruising (General disorders) | 6 (6) | 5 (6)
Injection site pain (General disorders) | 8 (10) | 1 (1)
COVID-19 (Infections and infestations) | 16 (16) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (7)
Sinusitis (Infections and infestations) | 8 (9) | 1 (1)
Palpatory finding abnormal (Investigations) | 11 (12) | 10 (11)
Weight increased (Investigations) | 2 (2) | 4 (4)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 6 (7)
Headache (Nervous system disorders) | 45 (61) | 18 (21)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT05386030/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT05386030/SAP_001.pdf